CLINICAL TRIAL: NCT04128982
Title: Evaluation of the Impact of Sellick's Manoeuvre or Para-tracheal Compression of the Cervical Esophagus on Laryngeal Mass Movement and Vocal Cord Visualization in Obese Patients.
Brief Title: Vidéolaryngoscopy Study of the LPEC in Obese Patients
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: LPECOBESITY
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Videolaryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Videolaryngoscopy: Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression in 2 groups: patient in dorsal decubitus or Rapid Airway Management Positioner.
  Interventions: Procedure: mobilization of the larynx

INTERVENTIONS:
Procedure: mobilization of the larynx — Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression in 2 groups: patient in dorsal decubitus or Rapid Airway Management Positioner.

SUMMARY:
1. Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression in obese patient
2. International surveys comparing tracheal intubation difficulty on a scale of 1 to 3 between cricoid pressure, Left Paratracheal Esophageal Compression and neutral position

DETAILED DESCRIPTION:
Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression in obese patient

International surveys comparing tracheal intubation difficulty on a scale of 1 to 3 between cricoid pressure, Left Paratracheal Esophageal Compression and neutral position

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with BMI > 35 undergoing general anaesthesia

Exclusion Criteria:

* pregnant women
* people with facial
* oropharyngeal abnormalities

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults patients obese
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Distance between oesophagus and trachea | During laryngoscopy
  Distance between oesophagus and trachea

CONTACTS AND LOCATIONS:
Locations (1):
- Javillier, Liège, Belgium